CLINICAL TRIAL: NCT06027918
Title: The Effect of Altitude Difference on the Duration of Infraclavicular Peripheral Block Applied to Patients With Hand and Forearm Fractures; a Three-center Study in Adults at 100, 675, 1726 Meters
Brief Title: The Effect of Altitude Difference on the Duration of Nerve Block; A Three-Center Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fatma Acil,MD, Principal Investigator, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 12.09.2022/266
Record Dates: First submitted 2023-08-29; First posted 2023-09-07 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Forearm Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group V (1726 meter altitude) (Active Comparator): In the application of infraclavicular brachial plexus blocks (coracoid approach); 1.5mg/kg dose of bupivacaine and 1mg/kg lidocaine mixture will be applied around the axillary artery in the 6 o'clock position under US guidance.
  The block will be applied only once, approximately 15-20 minutes before surgery.
  Interventions: Procedure: Infraclavicular brachial plexus block
- Group D (675 meter altitude) (Active Comparator): In the application of infraclavicular brachial plexus blocks (coracoid approach); 1.5mg/kg dose of bupivacaine and 1mg/kg lidocaine mixture will be applied around the axillary artery in the 6 o'clock position under US guidance.
  The block will be applied only once, approximately 15-20 minutes before surgery.
  Interventions: Procedure: Infraclavicular brachial plexus block
- Group H( 100 meter altitude) (Active Comparator): In the application of infraclavicular brachial plexus blocks (coracoid approach); 1.5mg/kg dose of bupivacaine and 1mg/kg lidocaine mixture will be applied around the axillary artery in the 6 o'clock position under US guidance.
  The block will be applied only once, approximately 15-20 minutes before surgery.
  Interventions: Procedure: Infraclavicular brachial plexus block

INTERVENTIONS:
Procedure: Infraclavicular brachial plexus block — In the application of infraclavicular brachial plexus blocks (coracoid approach); 1.5mg/kg dose of bupivacaine and 1mg/kg lidocaine mixture will be applied around the axillary artery in the 6 o'clock position under US guidance.

SUMMARY:
Infraclavicular brachial plexus block in hand and forearm surgery has the advantages of high success rate and low risk of complications and is useful in providing long-lasting and effective postoperative analgesia in these patients. In response to hypoxemia at high altitude, increased blood viscosity, decreased carbon monoxide diffusion capacity, increased cerebral arterial blood flow, decreased blood volume and decreased cardiac output occur. At high altitude, the serum level of local anesthetics may increase due to an increase in their ionized fraction and a decrease in their clearance. In this respect, the pharmacodynamic and pharmacokinetic properties of peripheral nerve blocks may be altered when performed at high altitude. The primary objective of this prospective study was to test the hypothesis that postoperative pain scores are higher in patients undergoing infraclavicular nerve block at high altitude than in patients at low altitude.

This multicenter prospective randomized study will be initiated after approval of the Ethics Committee of Health ScienceUniversity Diyarbakir Gazi Yasargil Training and Research Hospital. Patients will be recruited simultaneously in 3 hospitals, Hatay Training and Research Hospital, Hatay, Turkey (100 m above sea level);Health Science Health Science University Diyarbakir Gazi Yasargil Training and Research Hospital, Diyarbakir, Turkey (675 m above sea level) and Health Science University Van Regional and Training Research Hospital, Van, Turkey (1726 m above sea level).

Infraclavicular brachial plexus blocks (coracoid approach) will be performed by administering a local anesthetic mixture of 1.5 mg/kg lidocaine 2% + 1 mg/kg bupivacaine 0.5% at the 6 o'clock position of the axillary artery under US guidance.

DETAILED DESCRIPTION:
Group V (1726 meter altitude): In the application of infraclavicular brachial plexus blocks (coracoid approach); 1.5mg/kg dose of bupivacaine and 1mg/kg lidocaine mixture will be applied around the axillary artery in the 6 o'clock position under US guidance.

* The block will be applied only once, approximately 15-20 minutes before surgery.
* All patients will undergo electrocardiographic monitoring, oxygen saturation monitoring with pulse oximetry and blood pressure measurement with automatic pneumatic manometer before the application.
* Intravenous 1mg midazolam and 50 mcg fentanyl will be administered to all patients for premedication before the procedure.
* The amount of medication to be given to all patients will be prepared as 1.5mg/kg bupivacaine and 1mg/kg lidocaine.
* The prepared drug will be administered around the axillary artery at the appropriate anatomical location determined under ultrasound guidance.
* Ultrasound device will be used as a supportive device during the application.
* The application will be performed by an anesthesiologist with at least 5 years of experience.
* mode of delivery will be provided face to face and individually
* The administration will be only once, 20-30 minutes before the surgical procedure, with a dose adjustment of 1.5mg/kg bupivacaine and 1mg/kg lidocaine per kilogram of weight.
* The application will be made in the preoperative preparation room in the operating room of the hospital where the surgery will be performed.
* The local anesthetic dose to be used in the application will be calculated according to the weight of the patient. local anesthetics will be prepared by another anesthesiologist in the preoperative preparation room just before the application.
* In the postoperative period, if the pain intensity (VAS) is <4, 100 mg paracetamol will be administered intravenously, if VAS = 4, 100 mg tramadol will be administered intravenously

Group D (675 meter altitude): In the application of infraclavicular brachial plexus blocks (coracoid approach); 1.5 mg/kg dose of bupivacaine and 1mg/kg lidocaine mixture will be applied around the axillary artery in the 6 o'clock position under US guidance.

* The block will be applied only once, approximately 15-20 minutes before surgery.
* All patients will undergo electrocardiographic monitoring, oxygen saturation monitoring with pulse oximetry and blood pressure measurement with automatic pneumatic manometer before the application.
* Intravenous 1mg midazolam and 50 mcg fentanyl will be administered to all patients for premedication before the procedure.
* The amount of medication to be given to all patients will be prepared as 1.5 mg/kg bupivacaine and 1mg/kg lidocaine.
* The prepared drug will be administered around the axillary artery at the appropriate anatomical location determined under ultrasound guidance.
* Ultrasound device will be used as a supportive device during the application.
* The application will be performed by an anesthesiologist with at least 5 years of experience.
* mode of delivery will be provided face to face and individually
* The administration will be only once, 20-30 minutes before the surgical procedure, with a dose adjustment of 1.5 mg/kg bupivacaine and 1mg/kg lidocaine per kilogram of weight.
* The application will be made in the preoperative preparation room in the operating room of the hospital where the surgery will be performed.
* The local anesthetic dose to be used in the application will be calculated according to the weight of the patient. local anesthetics will be prepared by another anesthesiologist in the preoperative preparation room just before the application.
* In the postoperative period, if the pain intensity (VAS) is <4, 100 mg paracetamol will be administered intravenously, if VAS = 4, 100 mg tramadol will be administered intravenously

Comparator / control treatment Group H (100 meter altitude): In the application of infraclavicular brachial plexus blocks (coracoid approach); 1.5 mg/kg dose of bupivacaine and 1mg/kg lidocaine mixture will be applied around the axillary artery in the 6 o'clock position under US guidance.

* The block will be applied only once, approximately 15-20 minutes before surgery.
* All patients will undergo electrocardiographic monitoring, oxygen saturation monitoring with pulse oximetry and blood pressure measurement with automatic pneumatic manometer before the application.
* Intravenous 1mg midazolam and 50 mcg fentanyl will be administered to all patients for premedication before the procedure.
* The amount of medication to be given to all patients will be prepared as 1.5 mg/kg bupivacaine and 1 mg/kg lidocaine.
* The prepared drug will be administered around the axillary artery at the appropriate anatomical location determined under ultrasound guidance.
* Ultrasound device will be used as a supportive device during the application.
* The application will be performed by an anesthesiologist with at least 5 years of experience.
* mode of delivery will be provided face to face and individually
* The administration will be only once, 20-30 minutes before the surgical procedure, with a dose adjustment of 1.5 mg/kg bupivacaine and 1mg/kg lidocaine per kilogram of weight.
* The application will be made in the preoperative preparation room in the operating room of the hospital where the surgery will be performed.
* The local anesthetic dose to be used in the application will be calculated according to the weight of the patient. local anesthetics will be prepared by another anesthesiologist in the preoperative preparation room just before the application.
* In the postoperative period, if the pain intensity (VAS) is <4, 100 mg paracetamol will be administered intravenously, if VAS = 4, 100 mg tramadol will be administered intravenously

ELIGIBILITY:
Inclusion Criteria:

* Between 18-55 years old
* Body mass index between 20 and 25
* Patients with American Society of Anesthesiologists classification (ASA) physical status I or II

Exclusion Criteria:

* Patients aged younger than 18 and older than 55 years
* American Society of Anesthesiologists classification (ASA) ≥ III
* Body mass index (BMI) >35
* Known history of allergy to local anesthetics preoperative chronic pain and therefore long-term analgesic use
* In case of coagulopathy
* Have a condition that constitutes a contraindication for the application of the block (local infection, sepsis, local anesthetic medicine allergy; severe neurological, muscular or psychiatric disease, coagulation disorders)
* With marked cognitive impairment
* Patients who did not want to participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | will be evaluated at 0, 4th, 8th, 12th, 14th, 16th, 18th, 24th hours postoperatively
  * The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
  * Pain intensity at the site of the operation.

SECONDARY OUTCOMES:
total amount of intravenous analgesics consumed | will be evaluated at 0, 4th, 8th, 12th, 14th, 16th, 18th, 24th hours postoperatively
  to be evaluated at the end of 24 hours postoperatively
Sensory block start time | The sensory block will be evaluated approximately 10 minutes after the application. It will be observed up to a maximum of 30 minutes.
  The onset time of sensory block was defined as the time to reach an absence of hot-cold sensation in all 4 nerve distributions after completion of injection of the local anesthetic mixture.
  Sensory block was assessed using the cold test on the dermatomes of the median, ulnar, radial and musculocutaneous nerves. Sensory block was graded on a 3-point scale (0: normal sensation, 1: analgesia [patient can feel touch but not cold], 2: anesthesia [patient cannot even feel touch]).
sensory block end time | It will be evaluated every hour after the implementation, up to a maximum of 120 hours.
  Sensory block end time: defined as the time when the hot-cold sensation disappears in all 4 nerve distributions after the injection of the local anesthetic mixture is completed.
Time to onset of motor block | Motor block onset time will be assessed every 10 minutes after the intervention until 60 minutes.
  Time to onset of motor block, the time from the completion of injection of the local anesthetic mixture until complete motor block develops (in case of bromage : 4).
  Motor block was assessed with the Modified Bromage scale (scale 0: full flexion of the fingers, wrist and elbow; scale 1: full flexion of the fingers and wrist, but no flexion of the elbow); scale 2: full flexion of the fingers, but no flexion of the wrist and elbow; scale 3: complete motor block; no flexion of the fingers, wrist and elbow).
Motor block end time | It will be evaluated every hour after the implementation, up to a maximum of 120 hours.
  Motor block was assessed with the Modified Bromage scale (scale 0: full flexion of the fingers, wrist and elbow; scale 1: full flexion of the fingers and wrist, but no flexion of the elbow); scale 2: full flexion of the fingers, but no flexion of the wrist and elbow; scale 3: complete motor block; no flexion of the fingers, wrist and elbow).
  If the bromage is 0, the motor block will be considered as eliminated.

CONTACTS AND LOCATIONS:
Overall Officials: Cem K. Kaçar, Assoc.Prof, Study Director — Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Locations (1):
- Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Harmon D, Frizelle HP. Supraclavicular block for day-case anaesthesia at altitude. Anaesthesia. 2001 Feb;56(2):197. doi: 10.1046/j.1365-2044.2001.01870-30.x. No abstract available. PMID 11167511